CLINICAL TRIAL: NCT03609593
Title: A Single-arm, Multi-center Phase II Trial of Bendamustine/rituximab Induction Followed by Venetoclax and Rituximab Consolidation for the Frontline Treatment of Chronic Lymphocytic Leukemia (CLL)
Brief Title: Bendamustine/rituximab Followed by Venetoclax and Rituximab for Treatment of Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nicole Lamanna (Other)
Responsible Party: Sponsor-Investigator, Nicole Lamanna, Associate Clinical Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAR6357
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia (CLL); Leukemia; Bendamustine; Rituximab; Venetoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Bendamustine Hydrochloride; venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BR followed by venetoclax and rituximab (Experimental): Subjects will be on Bendamustine 50-90 mg/m2 on days 1-2 for three cycles with each cycle being 28 days, and Rituximab 375 mg/m2 on day 1 or days 1-2 for three cycles with each cycle being 28 days. Venetoclax will then be started in a step-wise fashion per the package insert.
  Interventions: Drug: Bendamustine; Drug: Venetoclax; Drug: Rituximab

INTERVENTIONS:
Drug: Bendamustine — Subjects will receive Bendamustine 50-90 mg/m2 on days 1-2 for three cycles with each cycle being 28 days.
  Other Names: Treanda
Drug: Venetoclax — Venetoclax: 12 cycles
  Venetoclax will then be started after 3 cycles of BR. Dosing for venetoclax will be in a step wise fashion as follows:
  * Cycle 4 days 1-7 (Week 1): 20 mg once daily
  * Cycle 4 days 8-14 (Week 2): 50 mg once daily
  * Cycle 4 days 15-21 (Week 3): 100 mg once daily
  * Cycle 4 days 22-28 (Week 4): 200 mg once daily
  * Cycle 4 day 29 and thereafter (Week 5 and on): 400 mg once daily; continue until disease progression, unacceptable toxicity, or 12 cycles duration.
  Other Names: ABT-199; Venclexta
Drug: Rituximab — For cycles 1 through 3, subjects will receive BR on days 1 and 2. For cycles 5-10, subjects will receive rituximab monotherapy at 375 mg/m2 (cycle 5) or rituximab at 500 mg/m2 (cycles 6-10) on day 1 (or days 1 and 2 if split-dose).
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine the efficacy of bendamustine and rituximab (BR) followed by venetoclax for 12 months. The total time on therapy is 15 months. Bendamustine and rituximab is a commonly used treatment for CLL. Venetoclax is an oral drug that blocks a protein called BCL-2 which is present on CLL cells. It is approved for patients with relapsed (the cancer has come back) or refractory (the cancer did not respond) CLL who harbor a deletion in the short arm of chromosome 17 [del(17p)]. When this drug is used by itself, many patients needed to be admitted to the hospital to monitor for a complication known as tumor lysis syndrome. This is an oncologic emergency that is caused by massive destruction of tumor cells with the release of large amounts of electrolytes and other molecules into the blood that can lead to renal failure and potentially death.

DETAILED DESCRIPTION:
This is a single arm multicenter phase II study using bendamustine-rituximab (BR) followed by venetoclax and rituximab for the upfront treatment of chronic lymphocytic leukemia (CLL). The activity, safety, and survival data have been presented previously for BR alone in patients with previously untreated disease and venetoclax alone in relapsed/refractory patients and those with high-risk disease. After pretreatment evaluation, patients will receive three cycles of BR followed by venetoclax via a five-week dose escalation to 400 mg daily. Once patients reach 400 mg of venetoclax daily, patients will receive six cycles (months) of rituximab as consolidation. Total time of venetoclax therapy will be 12 cycles and total time on therapy (BR plus venetoclax plus rituximab) will be 15 cycles. Responses and endpoints will be assessed after 3, 6, 9 (laboratory only), 12, 18, 24, 30, and 36 cycles. Minimal residual disease (MRD) testing will be done after 3, 6, 9, 12, 18, and 24 cycles via an 8-color flow cytometry panel. Bone marrow testing for MRD can be performed if the peripheral blood is MRD negative (or was MRD negative at the last test). Anti-infective prophylaxis against H. zoster and P. jiroveci will be mandated. Tumor lysis syndrome (TLS) prophylaxis with allopurinol and/or an alternative will be mandated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age.
* Diagnosed with CLL
* To be considered CLL, the subject must have an absolute lymphocytosis in the blood of at least 5,000 lymphocytes per microliter, or bone marrow lymphocytosis greater than or equal to 30% of all nucleated cells.
* Histologic and immunophenotypic analysis should demonstrate small to moderate size lymphocytes with flow cytometry demonstrating a certain population of lymphocytes.
* No prior therapy for their disease. Topical or inhaled corticosteroids are permitted for other medical conditions, ie asthma or dermatologic reasons.
* Eastern Oncology Cooperative Group (ECOG) performance score of ≤ 2.
* Subjects with autoimmune hemolytic anemia or autoimmune thrombocytopenia will be eligible for treatment on this protocol regardless of disease stage upon discussion with the principal investigator.
* An absolute neutrophil count > 1.0 109/L; hemoglobin > 8 g/dL; or a platelet count > 50 x 109/L (unless due to bone marrow failure).
* Adequate hepatic function
* activated partial thromboplastin time (aPTT) and prothrombin time (PT) not to exceed 1.5x the upper limit of reference ranges.
* Ability to understand and the willingness to sign a written informed consent document.
* Women of child-bearing potential and men must agree to use adequate contraception (see below) for at least 90 days prior to study entry and for the duration of study participation.

  * For women of childbearing potential (WCBP): a negative serum β-human chorionic gonadotropin (βhCG) pregnancy test must be performed within 1 week before randomization (WCBP defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally post-menopausal for at least 24 consecutive months [women ≤ 55 years] or 12 consecutive months [women > 55 years]).
  * Male and female subjects who are not surgically sterile or postmenopausal must be willing to use medically acceptable methods of birth control from the first dose of study drug to 30 days after the last dose of study drug. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception.

Exclusion Criteria:

* Subjects who have been previously treated for CLL or small lymphocytic lymphoma (SLL), except with corticosteroids for symptom relief.
* Treatment with any of the following within 7 days prior to the first dose of study drug:

  * Steroid therapy for anti-neoplastic intent
  * moderate or strong cytochrome P450 3A (CYP3A) inhibitors
  * moderate or strong CYP3A inducers
* Subject has known allergy to both xanthine oxidase inhibitors and/or rasburicase.
* Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study.
* Subject has evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  1. Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
  2. Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate.
* Subject is known to be positive for HIV. (HIV testing is not required.)
* New York Heart Association (NYHA) class II-IV heart failure or arrhythmia requiring treatment.
* Pregnant or lactating women. Women and men of childbearing age should use effective contraception.
* Subject has a history of active malignancies other than CLL within the past 2 years prior to study entry with the exception of: adequately treated in situ carcinoma of the cervix uteri, adequately treated basal cell carcinoma or localized squamous cell carcinoma of the skin, or previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Subjects may receive intravenous immunoglobulin (IVIG) for hypogammaglobulinemia while on protocol. Subjects may receive erythropoietin, filgrastim, pegfilgrastim, or sargramostim while on protocol.
* Subject has malabsorption syndrome or other condition that precludes enteral route of administration.
* Subjects with known Richter's syndrome or a history of Richter's syndrome.
* Subjects who are are actively being treated for a non-hematologic autoimmune disease, or are on other immunomodulatory agents (e.g. cyclosporine, tacrolimus, etc.) will be excluded.
* Subjects who have received an allogeneic stem cell transplant.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BCL-2 inhibitors, bendamustine, or anti-CD20 monoclonal antibodies.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * Grapefruit or grapefruit products
  * Seville oranges (including marmalade containing Seville oranges)
  * Star fruit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) after the completion of all therapy | 15 months
  Proportion of patients with reduction in tumor burden of a predefined amount

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Lamanna, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No